CLINICAL TRIAL: NCT05820295
Title: Improving How Older Adults at Risk for Cardiovascular Outcomes Are Selected for Care Coordination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-09025263; 1K18HS029255-01 (AHRQ)
Record Dates: First submitted 2023-04-07; First posted 2023-04-19 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases; Myocardial Infarction; Atrial Fibrillation; Diabetes Mellitus; Heart Failure; Hyperlipidemias; Hypertension; Ischemic Heart Disease; Stroke; Transient Ischemic Attack
Keywords: care coordination; accountable care organization
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Atrial Fibrillation; Diabetes Mellitus; Heart Failure; Hyperlipidemias; Hypertension; Myocardial Ischemia; Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will assign care coordinators to individuals based on perceived need for assistance with care coordination. Perceived need will be measured through a proxy's responses to a previously validated telephone survey on perceptions of care coordination.
  Interventions: Behavioral: Care coordination delivered based on perceived need
- Control (Active Comparator): Usual care assigns patients to care coordinators in response to a discharge from a hospital or a direct referral from a physician.
  Interventions: Behavioral: Care coordination delivered based on usual care (e.g. discharge from hospital)

INTERVENTIONS:
Behavioral: Care coordination delivered based on perceived need — If patients in intervention group report on the survey that they experience difficulty coordinating care among their providers, the patient will be selected for care management services. Those services will attempt to address the problems with care coordination that the proxy reported.
  Arms: Intervention
Behavioral: Care coordination delivered based on usual care (e.g. discharge from hospital) — If a patient is discharged from a hospital, the patient will be selected for care management services.
  Arms: Control

SUMMARY:
This pragmatic clinical trial embedded in an accountable care organization will determine the comparative effectiveness of two approaches for assigning care coordinators to older adults at risk for cardiovascular outcomes. The hypothesis is that assigning care coordinators to older adults based on perceived need will be more effective at preventing emergency department visits and hospitalizations compared to usual care.

DETAILED DESCRIPTION:
This project will use a pragmatic clinical trial embedded in an accountable care organization (ACO) to determine the comparative effectiveness of two different approaches for selecting older adults at risk for cardiovascular outcomes to receive support from care coordinators: (1) an approach that assigns older adults to care coordinators based on self-reported difficulty with care coordination, or (2) usual care, which generally assigns older adults to care coordinators after hospital discharge, regardless of perceived need. The investigators will include community-dwelling Medicare beneficiaries ≥65 years old with cardiovascular disease (CVD) or 1 or more CVD risk factors who have been attributed to the NewYork Quality Care ACO and who have fragmented care. The investigators will randomize the participants into two groups. This study is highly pragmatic, and the intervention is sustainable and scalable. Moreover, the proposed approach has the potential to improve care delivery and outcomes for older adults at risk for cardiovascular outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Medicare beneficiaries 65 years and older,
* Attributed to the NewYork Quality Care accountable care organization,
* Are community-dwelling,
* Have cardiovascular disease or 1 or more cardiovascular risk factors, and
* Had highly fragmented ambulatory care in the prior year (defined as a reversed Bice-Boxerman Index greater than or equal to 0.85)

Exclusion Criteria:

* Those who reside in long-term care or nursing home facilities (based on addresses in Medicare claims)
* Enrolled in home hospice
* Dementia (as measured in claims using the Bynum Standard 1-year definition)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Kern, MD, MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital - Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 202 | 198
Completed | 202 | 198
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 202 | 198 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.1 (7.1) | 75.8 (7.0) | 75.8 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 146 | 287
  Male | 61 | 52 | 113
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 143 | 141 | 284
  Non-white | 59 | 57 | 116
Enrollment type [Count of Participants; unit: Participants] — Reason for enrollment in Medicare
  Participants
    65 years and older, and dually eligible for Medicaid | 69 | 67 | 136
    65 years and older, not dually eligible for Medicaid | 132 | 131 | 263
    End-stage renal disease | 1 | 0 | 1
    Disability | 0 | 0 | 0
Co-morbidities [Count of Participants; unit: Participants]
  Acute myocardial infarction | 0 | 3 | 3
  Atrial fibrillation | 19 | 28 | 47
  Chronic kidney disease (not end-stage) | 35 | 34 | 69
  Chronic obstructive pulmonary disease and bronchiectasis | 19 | 37 | 56
  Colorectal cancer | 9 | 4 | 13
  Depression | 43 | 44 | 87
  Diabetes | 64 | 60 | 124
  Endometrial cancer | 2 | 6 | 8
  End-stage renal disease | 1 | 3 | 4
  Female or male breast cancer | 25 | 25 | 50
  Heart failure | 29 | 30 | 59
  Hyperlipidemia | 162 | 159 | 321
  Hypertension | 154 | 143 | 297
  Ischemic heart disease | 71 | 82 | 153
  Lung cancer | 7 | 4 | 11
  Prostate cancer | 13 | 13 | 26
  Stroke / transient ischemic attack | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Emergency Department Visits or Hospital Admissions
Description: Occurrence of an emergency department visit or hospital admission, as measured in Medicare claims. This outcome measure allows more than one event per participant.
Time Frame: Over 12 months (beginning 1 month after the start of care coordination)
Measure: Number (95% Confidence Interval); unit: events per 100 person-days alive
Arm/Group | Intervention | Control
Number analyzed (Participants) | 202 | 198
events per 100 person-days alive | 0.25 [0.21 to 0.31] | 0.21 [0.17 to 0.27]

2. Secondary Outcome: Acceptability
Description: Number of people in each group who accept care management
Time Frame: Up to 1 year of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 202 | 198
Participants | 13 | 17

3. Secondary Outcome: Appropriateness
Description: Number of participants who requested care management services that were in scope for the care managers' credentials
Time Frame: Up to 1 year of follow-up
Population: This outcome is restricted to those who accepted care management.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 13 | 17
Participants | 13 | 17

4. Secondary Outcome: Fidelity
Description: Number of participants who received care management services, among those who requested care management services.
Time Frame: Up to 1 year of follow-up
Population: This measure is restricted to those who requested care management services.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 13 | 17
Participants | 13 | 17

5. Secondary Outcome: Efficiency
Description: The total number of care management encounters per group. This measure allows more than one encounter per participant.
Time Frame: Up to 1 year of follow-up
Measure: Number; unit: Encounters
Arm/Group | Intervention | Control
Number analyzed (Participants) | 202 | 198
Encounters | 52 | 45

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 4/202 | 1/198
Serious Adverse Events (participants affected / at risk) | 0/202 | 0/198
Other Adverse Events (participants affected / at risk) | 0/202 | 0/198

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT05820295/Prot_SAP_000.pdf